CLINICAL TRIAL: NCT01986504
Title: The Johns Hopkins Transplant Infectious Diseases Prospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Kieren Marr, Professor of Medicine, Johns Hopkins University
Other Study IDs: NA_00044645
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Transplantation
Keywords: Infection; Cohort; Prospective; Epidemiology; Outcome
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The Transplant Infectious Diseases Prospective Cohort Study facilitates the prospective identification and collection of data of infectious disease complications in order to determine the epidemiology, risk factors, and outcomes of patients who receive solid organ or stem cell or plastic surgery transplants at Johns Hopkins and other transplant centers. It is essential for the care and treatment of this population to employ a mechanism for investigators to centralize these datasets, using standardized definitions of infectious complications. This protocol outlines the procedures to be utilized in order to prospectively follow the diagnosis and treatment of infectious complications in transplant patients.

DETAILED DESCRIPTION:
Patients are approached at their transplant screening visit, if possible, or during their hospital stay (before or after transplant) in order to introduce the study and obtain informed consent for participation. A letter to transplant physicians will introduce this study. Data collection will begin immediately upon consent and continue for up to five years. The informed consent form specifically requests permission to contact the subject in the future to verify information or if the subject is lost to follow up by Transplant services.

The Day of transplant will be considered day 0 for enrollment in this observational study. Data will be collected on clinical template forms completed by study team members, as infectious complications become apparent in either outpatient ID clinics or on the inpatient service. A member of the research team will complete data collection in the registry, maintained on the REDCap platform. In addition, patient electronic records will be reviewed every 3 months to identify and record infectious complications, treatments administered, and outcomes. During these intervals, subjects will be contacted by phone to review the same outcomes.

Creation of the registry relies on use of standardized definitions to define infections. An electronic database has been constructed in the REDCap system, documenting subject demographics, transplant variables, infection variables, treatments administered, and overall outcomes, during each interim time period.

ELIGIBILITY:
Inclusion Criteria:

Hematopoietic stem cell (bone marrow) and solid organ transplant patients -

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hematopoietic stem cell (bone marrow) and solid organ transplant patients
Sampling Method: Probability Sample
Enrollment: 1058 (Actual)
Dates: Start 2011-06; Primary Completion 2014-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Epidemiology and Outcomes | 6 years
  This protocol will enable the creation of a prospective registry of infectious complications in transplant patients, to be used for research epidemiology and outcomes, and, ultimately, to improve patient care.

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States